CLINICAL TRIAL: NCT06841107
Title: Investigation of the Effect of Spine Health Training and Lumbar Region Support on Back Pain and Discomfort in City Bus Drivers: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Ece Arık, Principal Investigator, Pamukkale University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: E-60116787-020-244556
Record Dates: First submitted 2025-01-25; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Low Back Pain (LBP); Low Back Disorder
Keywords: Lumbar Region Support
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: 1. group was given training on spinal health.
  2. group was given lumbar region support along with training on spine health.
  3. group (control group) received no intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Spinal health training (Active Comparator): It focuses on basic body knowledge, correct posture and spinal health; common spinal problems, especially in drivers, and their prevention. It covers how a healthy spine should look like, what to look out for during and after working hours, correct driver seat adjustments and stretching and strengthening exercises to maintain spinal health.
  Interventions: Other: Training was provided on spinal health.
- Spinal health training and lumbar region support (Active Comparator): It focuses on basic body knowledge, correct posture and spinal health; common spinal problems, especially in drivers, and their prevention. It covers how a healthy spine should look like, what to look out for during and after working hours, correct driver seat adjustments and stretching and strengthening exercises to maintain spinal health. In addition, lumbar region support was used during working hours for 3 months.
  Interventions: Other: Training on spinal health was provided and lumbar region support was applied for 3 months.
- Control (No Intervention): Control group; there is no intervention.

INTERVENTIONS:
Other: Training was provided on spinal health. — Bus drivers were told about the practices they could do during and outside of work hours, and were asked to comply with these practices every day for 3 months.
  Arms: Spinal health training
Other: Training on spinal health was provided and lumbar region support was applied for 3 months. — Bus drivers were told about the practices they could do during and outside of work hours, and were asked to comply with these practices every day for 3 months. In addition, lumbar region support was used every day during working hours for 3 months.
  Arms: Spinal health training and lumbar region support

SUMMARY:
The World Health Organization (WHO) classifies driving as a function of daily activities and social participation. Professional bus drivers have an important place in society for transportation. Drivers are seen as a stressful occupational group due to their use of the vehicle in the same position and intensive working hours.

It is important for bus drivers not to feel discomfort during long working hours and to choose the right seat position. Because the design of the driver's seat directly affects the driver's spine biomechanics. For an ergonomic posture, the head, back and waist areas of the driver's seats should be well supported. During driving, the waist and back of the seat should be supported in order to fix the driver's lumbar region due to movements in the vehicle seat.

Professional drivers' long working hours, sitting positions and exposure to vibration, work stress, short breaks, and insufficient physical activity bring about occupational diseases. Musculoskeletal disorders are seen primarily, as well as hypertension, diabetes, cardiovascular diseases, etc. Most musculoskeletal problems are caused by incorrect sitting positions. In many studies, it is seen that drivers have neck, upper back and waist pain, and spinal problems. The main reason for musculoskeletal disorders is that the seats are not adjustable and most drivers try to maintain their posture with additional supports. When the studies conducted look at the relationship between the driver and the seat during long-term vehicle use, the pressure in the contact areas, insufficient support in the back and waist area causes a decrease in comfort, thus causing back and waist discomfort and pain in the individual.

Psychosocial factors are also risk factors affecting musculoskeletal disorders. It has been observed that stress causes various diseases including heart disease, gastrointestinal diseases, and musculoskeletal disorders in city bus drivers. Psychosocial factors such as job satisfaction, burnout, and stress have been found to be associated with the incidence of musculoskeletal disorders.

Eliminating the back pain and discomfort of professional drivers, who occupy a large place in society, will provide great benefits both for the health of individuals and to alleviate the burden on the service sector. In studies in the international literature on this subject, only posture analyses of drivers have been conducted or the effects on pain and discomfort in the short term after the intervention have been examined. In the literature, drivers stated that seats with lumbo-sacral support were more comfortable than standard seats. In this study, the effect on pain and discomfort will be examined by following the drivers for 3 months. The aim of this study is to examine the effectiveness of the use of lumbar region support in bus drivers by following them for 3 months in terms of back pain and discomfort caused by long working hours and incorrect posture.

ELIGIBILITY:
Inclusion Criteria:

* Those with back pain and discomfort
* Those who have been a bus driver for at least 1 year

Exclusion Criteria:

* Having been a bus driver for less than 1 year
* Having any orthopedic, neurological, rheumatological or metabolic disease diagnosed due to back pain
* Having had spinal surgery
* Using medication for a diagnosed back problem
* Having received physiotherapy/physical therapy for a diagnosed back pain problem

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
The Rapid Entire Body Assessment (REBA) | 3 months
  Posture assessment was performed before the intervention and after three months of lumbar support use.
  The Rapid Entire Body Assessment (REBA) assesses the risk of musculoskeletal disorders by analyzing body posture during work. It rates the level of risk on a scale of 1 to 15, with higher scores indicating a higher risk of musculoskeletal disorders due to poor posture. This assessment was used to demonstrate the impact of posture on low back pain and discomfort.
Extended Nordic Musculoskeletal Questionnaire | 3 months
  A musculoskeletal questionnaire was conducted before the intervention and 3 months after the spine health training. The Extended Nordic Musculoskeletal Questionnaire was used to assess musculoskeletal disorders. This questionnaire collects information about current, past month and past 12 months musculoskeletal problems in nine different parts of the body (neck, shoulder, elbow, hand/wrist, back, waist, hip/thigh, knee, foot/ankle). It also collects information on how often these pains/discomforts occur, whether they decrease on vacation days and the severity of the pain. This questionnaire was used to evaluate the effectiveness of spine health training.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Kitiş, Professor, Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)